CLINICAL TRIAL: NCT00858780
Title: Dose Reduction or Discontinuation of Etanercept in Methotrexate-Treated Rheumatoid Arthritis Subjects Who Have Achieved a Stable Low Disease Activity-state (DOSERA)
Brief Title: Study Comparing The Effect On Disease Activity When Reducing Or Discontinuing Etanercept In Subjects With RA
Acronym: DOSERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0881K1-4500; B1801016
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 50mg once weekly + methotrexate
  Interventions: Drug: Etanercept
- 2 (Active Comparator): 25mg once weekly + methotrexate
  Interventions: Drug: Etanercept
- 3 (Placebo Comparator): once weekly + methotrexate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — 50 mg etanercept once weekly + methotrexate
  Arms: 1
Drug: Etanercept — 25mg etanercept once weekly + methotrexate
  Arms: 2
Drug: Placebo — Placebo comparator once weekly + methotrexate
  Arms: 3

SUMMARY:
This study involves Rheumatoid Arthritis patients in regular clinical setting who are already on etanercept treatment and are in remission or in a low disease activity (LDA) state, and is intended to identify parameters that can serve as guidance in clinical settings. This study will consider the clinical and radiographic course in subjects when etanercept treatment is tapered or discontinued, and analyze the subjects' experience of disease worsening and the predictive values of clinical parameters, serum biomarkers and imaging on the clinical and radiographic course in different treatment groups. The effect of re-treatment with etanercept at treatment failure will also be studied.

ELIGIBILITY:
Inclusion criteria:

* Subject has a current DAS28 equal to or less than 3.2.
* Subject is currently receiving treatment with etanercept, either 25 mg twice weekly or 50 mg once weekly, for a minimum of 14 months at baseline
* Subject is currently receiving oral, sc or intramuscular methotrexate once weekly, 7.5 mg/week to 25 mg/week and at a stable dose for a minimum of 4 months at baseline.

Exclusion Criteria:

* Subject has earlier had an attempt of discontinuing etanercept for reasons of remission or low disease activity state.
* Subject has received any disease-modifying anti-rheumatic drug, other than methotrexate, within one month before baseline.
* Subject has had a dose of prednisone (or equivalent) >7.5 mg/day or has received intra-articular, intravenous, intramuscular, or subcutaneous corticosteroid within one month of baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- Denmark (2):
  - Pfizer Investigational Site, Glostrup Municipality
  - Pfizer Investigational Site, Hellerup
- Finland (2):
  - Pfizer Investigational Site, Jyväskylä, Finland
  - Pfizer Investigational Site, Helsinki
- Hungary (3):
  - Pfizer Investigational Site, Gyula
  - Pfizer Investigational Site, Szombathely
  - Pfizer Investigational Site, Veszprém
- Pfizer Investigational Site, Reykjavik, Iceland
- Norway (3):
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Lillehammer
  - Pfizer Investigational Site, Oslo
- Sweden (4):
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uppsala

REFERENCES:
- [Derived] van Vollenhoven RF, Ostergaard M, Leirisalo-Repo M, Uhlig T, Jansson M, Larsson E, Brock F, Franck-Larsson K. Full dose, reduced dose or discontinuation of etanercept in rheumatoid arthritis. Ann Rheum Dis. 2016 Jan;75(1):52-8. doi: 10.1136/annrheumdis-2014-205726. Epub 2015 Apr 14. PMID 25873634
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881K1-4500&StudyName=Study%20Comparing%20The%20Effect%20On%20Disease%20Activity%20When%20Reducing%20Or%20Discontinuing%20Etanercept%20In%20Subjects%20With%20RA

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept 50 mg - Period 1: Etanercept 50 milligram (mg) subcutaneous (SC) injection once weekly along with methotrexate (MTX) 7.5 mg/week to 25 mg/week as a single dose or divided doses, as oral tablet or as SC or intramuscular (IM) injection, depending on the dose a participant was receiving at time of screening, for 8 weeks. Participants who maintained disease activity score based on 28-joints count (DAS28) less than or equal to (<=) 3.2 in Period 1 were randomized in Period 2.
- Etanercept 50 mg - Period 2: Etanercept 50 mg SC injection once weekly along with MTX 7.5 mg/week to 25 mg/week as a single dose or divided doses, as oral tablet or as SC or IM injection up to treatment failure or Week 48/early termination. Participants who showed treatment failure (DAS28 more than [>] 5.1, or DAS28 >3.2 but <=5.1 along with an increase from baseline in DAS28 more than or equal to [>=] 1.2, or DAS28 >3.2 along with an increase from baseline >=0.6 but <1.2 on 2 consecutive visits, or disease progression as determined by investigator) were reassigned to Period 3.
- Etanercept 25 mg - Period 2: Etanercept 25 mg SC injection once weekly along with MTX 7.5 mg/week to 25 mg/week as a single dose or divided doses, as oral tablet or as SC or IM injection up to treatment failure or Week 48/early termination. Participants who showed treatment failure (DAS28 >5.1 or DAS28 >3.2 but <=5.1 along with an increase from baseline in DAS28 >=1.2 or DAS28 >3.2 along with an increase from baseline >=0.6 but <1.2 on 2 consecutive visits or disease progression as determined by investigator) were reassigned to Period 3.
- Placebo - Period 2: Placebo matched to etanercept SC injection once weekly along with MTX 7.5 mg/week to 25 mg/week as a single dose or divided doses, as oral tablet or as SC or IM injection up to treatment failure or Week 48/early termination. Participants who showed treatment failure (DAS28 >5.1 or DAS28 >3.2 but <=5.1 along with an increase from baseline in DAS28 >=1.2 or DAS28 >3.2 along with an increase from baseline >=0.6 but <1.2 on 2 consecutive visits or disease progression as determined by investigator) were reassigned to Period 3.
- Etanercept 50 mg - Period 3: Participants, who showed treatment failure in Period 2, received etanercept 50 mg SC injection once weekly along with MTX 7.5 mg/week to 25 mg/week as a single dose or divided doses, as oral tablet or as SC or IM injection up to Week 48/early termination.
Period: Open-Label (OL) Run-In(Week-8 to Week 0)
Arm/Group | Etanercept 50 mg - Period 1 | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2 | Etanercept 50 mg - Period 3
Started | 91 | 0 | 0 | 0 | 0
Completed | 73 | 0 | 0 | 0 | 0
Not Completed | 18 | 0 | 0 | 0 | 0
Not completed — Did not enter double-blind period | 18 | 0 | 0 | 0 | 0
Period: Double-Blind (Week 0 to Failure/Week 48)
Arm/Group | Etanercept 50 mg - Period 1 | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2 | Etanercept 50 mg - Period 3
Started | 0 | 23 | 27 | 23 | 0
Completed | 0 | 21 | 25 | 22 | 0
Not Completed | 0 | 2 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0
Period: OL Re-Treatment (Failure to Week 48)
Arm/Group | Etanercept 50 mg - Period 1 | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2 | Etanercept 50 mg - Period 3
Started | 0 | 0 | 0 | 0 | 43 (43 participants showed treatment failure in Period 2 and entered in Period 3.)
Completed | 0 | 0 | 0 | 0 | 41
Not Completed | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants who were enrolled in this study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 91
Age Continuous [Mean (Standard Deviation); unit: years] | 56.14 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participant Who Were Non-Failures
Description: A participant was considered as non-failure if the calculated DAS28 <=3.2 at all visits or if the calculated DAS28 >3.2, the increase of calculated DAS28 from randomization (Week 0): was <0.6 at all visit or was >=0.6 but <1.2 on no more than 1 consecutive visit. Percentage of participants who were non-failures calculated based on DAS28 and disease progression as determined by investigator or participant.
Time Frame: Week 48
Population: Modified intent-to-treat (m-ITT) analysis set included all randomized participants who received at least 1 dose of study medication after randomization and had at least 1 available evaluation after the first administration of study medication after randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
percentage of participants | 52.2 | 44.4 | 13.0
Statistical Analysis 1: Comparison: Etanercept 50 mg - Period 2 vs Placebo - Period 2; Analysis was performed using a generalized estimating equations (GEE) model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment groups, visits, their interaction, and the stratification factor as factors in the model; Test type: Superiority or Other; p = 0.007, GEE Model; Odds Ratio (OR) = 7.17, 95% CI 2-sided [1.72 to 29.82]
Statistical Analysis 2: Comparison: Etanercept 50 mg - Period 2 vs Etanercept 25 mg - Period 2; Analysis was performed using a GEE model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment groups, visits, their interaction, and the stratification factor as factors in the model; Test type: Superiority or Other; p = 0.362, GEE Model; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.54 to 5.41]
Statistical Analysis 3: Comparison: Etanercept 25 mg - Period 2 vs Placebo - Period 2; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.044, GEE Model; Odds Ratio (OR) = 4.20, 95% CI 2-sided [1.04 to 16.99]

2. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF (in weeks): (date of failure minus date of randomization) divided by 7. Date of failure was ordinary visit date or extra visit date in case of failure (extra visit was within 2 weeks from the date a participant experienced significant disease progression between visits and wanted to withdraw from Period 2), or date of withdrawal due to disease progression. Participants who did not have a treatment failure were censored at their last evaluation visit. Participants who withdrew from the study prematurely and did not have a treatment failure were censored on the date of their withdrawal.
Time Frame: Randomization (Week 0) up to date of failure, withdrawal due to disease progression or last evaluation visit (Week 48)
Population: m-ITT analysis set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
weeks | 48.0 [18.1 to NA] — Upper limit of confidence interval was not evaluable since there were only 50% treatment failures and there was lack of information on the later failure times. | 36.1 [15.6 to NA] — Upper limit of confidence interval was not evaluable since there were only 50% treatment failures and there was lack of information on the later failure times. | 6.1 [4.0 to 8.4]

3. Secondary Outcome: Percentage of Participants With Remission or Low Disease Activity (LDA)
Description: Participants who had DAS28 less than or equal to (<=) 3.2 were considered in remission or LDA state.
Time Frame: Baseline (Week -8), Week -4, Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: m-ITT analysis set. Here, 'n' signifies participants evaluable for each time-point for each treatment arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
percentage of participants
  Baseline (n= 19, 23, 19) | 100 | 100 | 100
  Week -4 (n= 23, 26, 23) | 100 | 100 | 100
  Randomization (n= 22, 27, 23) | 100 | 96.3 | 100
  Week 6 (n= 21, 26, 15) | 90.5 | 80.8 | 60.0
  Week 12 (n= 18, 21, 6) | 94.4 | 85.7 | 83.3
  Week 18 (n= 16, 19, 3) | 87.5 | 89.5 | 100
  Week 24 (n= 14, 16, 3) | 100 | 100 | 100
  Week 30 (n= 14, 15, 3) | 92.9 | 100 | 66.7
  Week 36 (n= 13, 14, 2) | 100 | 85.7 | 100
  Week 42 (n= 12, 12, 2) | 100 | 100 | 100
  Week 48 (n= 12, 12, 2) | 83.3 | 91.7 | 100

4. Secondary Outcome: Percentage of Visits During Which Participants Were in Remission or Low Disease Activity State
Description: Participants who had DAS28 <=3.2 were considered in remission or LDA state. Percentage of visits during which a participant was in remission or LDA state was calculated as number of visits in which participant was in remission or LDA divided by total number of visits multiplied by 100.
Time Frame: Randomization (Week 0) up to Week 48
Population: m-ITT analysis set. Here, N (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: percentage of visits
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 22 | 27 | 15
percentage of visits | 82.7 (31.1) | 74.8 (38.0) | 55.3 (48.5)

5. Secondary Outcome: Disease Activity Score Based on 28-Joint Count (DAS28) at Randomization
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PtGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 <=3.2 implied low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity and less than (<) 2.6=remission.
Time Frame: Randomization (Week 0)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 22 | 27 | 23
units on a scale | 1.86 (0.62) | 1.93 (0.85) | 1.93 (0.71)

6. Secondary Outcome: Change From Randomization in Disease Activity Score Based on 28-Joint Count (DAS28) at Week 6, 12, 18, 24, 30, 36, 42, and 48
Description: DAS28 calculated from SJC and PJC using the 28 joints count, the ESR (mm/hour) and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 <=3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity and <2.6=remission.
Time Frame: Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 21 | 26 | 15
units on a scale
  Change at Week 6 | 0.11 (0.24) | 0.47 (0.25) | 0.85 (0.36)
  Change at Week 12 | 0.38 (0.25) | 0.32 (0.26) | 1.33 (0.53)
  Change at Week 18 | 0.41 (0.25) | 0.64 (0.27) | 1.14 (0.69)
  Change at Week 24 | -0.00 (0.26) | 0.66 (0.28) | 1.02 (0.69)
  Change at Week 30 | 0.24 (0.26) | 0.74 (0.28) | 1.12 (0.69)
  Change at Week 36 | 0.18 (0.26) | 1.00 (0.28) | 0.45 (0.80)
  Change at Week 42 | 0.14 (0.27) | 0.45 (0.29) | 1.02 (0.80)
  Change at Week 48 | 0.46 (0.27) | 0.92 (0.29) | 1.17 (0.80)

7. Secondary Outcome: Change From Randomization in Tender Joints Count (TJC) at Week 6, 12, 18, 24, 30, 36, 42, and 48
Description: Number of tender joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1. A negative value in change from randomization indicates an improvement.
Time Frame: Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: m-ITT analysis set. Here, 'n' signifies participants evaluable for each time point for each treatment arm, respectively.
Measure: Median (Full Range); unit: tender joints
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
tender joints
  Randomization (n=23,27,23) | 0.0 [0 to 2] | 0.0 [0 to 2] | 0.0 [0 to 3]
  Change at Week 6 (n= 22, 26, 15) | 0.0 [-2 to 6] | 0.0 [-2 to 9] | 1.0 [0 to 9]
  Change at Week 12 (n= 18, 21, 6) | 0.0 [0 to 6] | 0.0 [-2 to 2] | 0.5 [0 to 24]
  Change at Week 18 (n= 16, 19, 3) | 0.0 [-1 to 2] | 0.0 [-2 to 6] | 0.0 [0 to 0]
  Change at Week 24 (n= 14, 16, 3) | 0.0 [0 to 0] | 0.0 [-1 to 2] | 0.0 [0 to 1]
  Change at Week 30 (n= 14, 15, 3) | 0.0 [-1 to 7] | 0.0 [-2 to 7] | 0.0 [-1 to 4]
  Change at Week 36 (n= 13, 14, 2) | 0.0 [0 to 1] | 0.0 [-2 to 4] | -0.5 [-1 to 0]
  Change at Week 42 (n= 12, 12, 2) | 0.0 [-2 to 1] | 0.0 [-2 to 0] | -0.5 [-1 to 0]
  Change at Week 48 (n= 12, 12, 2) | 0.0 [-2 to 1] | 0.0 [-1 to 2] | 0.5 [0 to 1]

8. Secondary Outcome: Change From Randomization in Swollen Joints Count (SJC) at Week 6, 12, 18, 24, 30, 36, 42, and 48
Description: Number of swollen joints was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1. A negative value in change from randomization indicates an improvement.
Time Frame: Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: m-ITT analysis set. Here, 'n' signifies participants evaluable for each time point for each treatment arm, respectively.
Measure: Median (Full Range); unit: swollen joints
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
swollen joints
  Randomization (n=23,27,23) | 0.0 [0 to 3] | 0.0 [0 to 3] | 0.0 [0 to 1]
  Change at Week 6 (n= 22, 26, 15) | 0.0 [-1 to 5] | 0.0 [-1 to 11] | 0.0 [0 to 6]
  Change at Week 12 (n= 18, 21, 6) | 0.0 [-1 to 4] | 0.0 [-1 to 3] | 1.0 [0 to 6]
  Change at Week 18 (n= 16, 19, 3) | 0.0 [-1 to 2] | 0.0 [-3 to 8] | 0.0 [0 to 2]
  Change at Week 24 (n= 14, 16, 3) | 0.0 [-3 to 1] | 0.0 [-1 to 1] | 0.0 [0 to 1]
  Change at Week 30 (n= 14, 15, 3) | 0.0 [-2 to 5] | 0.0 [-3 to 3] | 0.0 [0 to 4]
  Change at Week 36 (n= 13, 14, 2) | 0.0 [-2 to 1] | 0.0 [-1 to 3] | 0.0 [0 to 0]
  Change at Week 42 (n= 12, 12, 2) | 0.0 [-1 to 3] | 0.0 [-1 to 1] | 0.0 [0 to 0]
  Change at Week 48 (n= 12, 12, 2) | 0.0 [-2 to 1] | 0.0 [-2 to 0] | 0.5 [0 to 1]

9. Secondary Outcome: Change From Randomization in Physician Global Assessment (PGA) of Disease Activity at Week 6, 12, 18, 24, 30, 36, 42, and 48
Description: PGA of disease activity was measured on a 0 to 100 millimeter (mm) Visual Analog Scale (VAS), with 0 mm = no disease activity and 100 mm = extreme disease activity.
Time Frame: Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: m-ITT analysis set. Here, N (number of participants analyzed) signifies participants who were evaluable for this measure and 'n' signifies participants evaluable for each time point for each treatment arm, respectively.
Measure: Median (Full Range); unit: mm
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 22
mm
  Randomization (n=23,27,22) | 4.00 [0.0 to 13.0] | 3.00 [0.0 to 30.5] | 2.25 [0.0 to 19.0]
  Change at Week 6 (n= 22, 26, 14) | 1.50 [-8.0 to 20.5] | 0.25 [-7.0 to 58.0] | 4.00 [-9.0 to 50.0]
  Change at Week 12 (n= 18, 21, 6) | 1.00 [-6.0 to 17.0] | 0.50 [-7.0 to 14.0] | 6.75 [-4.5 to 42.0]
  Change at Week 18 (n= 16, 19, 3) | 2.50 [-11.0 to 18.0] | 4.00 [-7.0 to 32.0] | 10.00 [-4.0 to 16.0]
  Change at Week 24 (n= 14, 15, 3) | 1.00 [-9.0 to 8.0] | 2.00 [-7.0 to 23.0] | 8.00 [-5.0 to 14.0]
  Change at Week 30 (n= 14, 15, 3) | 1.00 [-3.0 to 55.0] | 0.00 [-7.0 to 35.0] | 5.00 [-5.0 to 18.0]
  Change at Week 36 (n= 13, 14, 2) | 0.00 [-4.0 to 9.0] | 0.00 [-7.5 to 36.0] | -6.50 [-16.0 to 3.0]
  Change at Week 42 (n= 12, 12, 2) | 0.25 [-6.0 to 26.0] | -1.00 [-9.0 to 3.0] | -3.00 [-6.0 to 0.0]
  Change at Week 48 (n= 12, 12, 2) | 0.25 [-3.0 to 16.0] | -1.75 [-8.5 to 4.0] | -1.50 [-3.0 to 0.0]

10. Secondary Outcome: Change From Randomization in Participant Global Assessment (PtGA) of Disease Activity at Week 6, 12, 18, 24, 30, 36, 42, and 48
Description: Participants assessed the overall activity of their rheumatoid arthritis (RA) on a 0 to 100 mm VAS, where 0 mm = no disease activity and 100 mm = extreme disease activity.
Time Frame: Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: m-ITT analysis set. Here, 'n' signifies participants evaluable for each time point for each treatment arm, respectively.
Measure: Median (Full Range); unit: mm
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
mm
  Randomization (n=23,27,23) | 8.00 [0.0 to 72.0] | 12.00 [0.0 to 52.5] | 13.00 [0.0 to 41.0]
  Change at Week 6 (n= 22, 26, 15) | 2.50 [-20.0 to 42.5] | 0.25 [-25.5 to 57.0] | 10.00 [-33.0 to 57.0]
  Change at Week 12 (n= 18, 21, 6) | -0.25 [-18.5 to 16.0] | 0.00 [-15.0 to 28.0] | 18.00 [-28.0 to 51.0]
  Change at Week 18 (n= 16, 19, 3) | 0.00 [-18.5 to 62.0] | -0.50 [-9.5 to 26.0] | 20.00 [-27.0 to 21.0]
  Change at Week 24 (n= 14, 16, 3) | 0.00 [-22.5 to 10.0] | 0.50 [-18.5 to 27.0] | 4.00 [-22.0 to 11.0]
  Change at Week 30 (n= 14, 15, 3) | -1.00 [-22.5 to 47.0] | 0.50 [-29.5 to 9.5] | -5.50 [-27.0 to 38.5]
  Change at Week 36 (n= 13, 14, 2) | 0.00 [-24.5 to 13.0] | 0.50 [-9.5 to 16.5] | -24.00 [-38.0 to -10.0]
  Change at Week 42 (n= 12, 12, 2) | -0.50 [-21.5 to 29.0] | -0.25 [-28.5 to 27.0] | -7.50 [-27.0 to 12.0]
  Change at Week 48 (n= 12, 12, 2) | 1.50 [-24.0 to 22.0] | -1.00 [-34.5 to 12.0] | -7.00 [-26.0 to 12.0]

11. Secondary Outcome: Participant General Health Visual Analog Scale (VAS) at Randomization
Description: Participants answered "in general how would you rate your health over the last 2-3 weeks?" Participants responded by using a 0 to 100 mm VAS, where 0 mm = very well and 100 mm = extremely bad.
Time Frame: Randomization (Week 0)
Population: m-ITT analysis set.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
mm | 14.43 (12.87) | 15.11 (13.15) | 18.52 (15.35)

12. Secondary Outcome: Change From Randomization in Participant General Health Visual Analog Scale (VAS) at Week 6, 12, 18, 24, 30, 36, 42, and 48
Description: as for outcome 11
Time Frame: Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: m-ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
mm
  Change at Week 6 | 8.21 (4.74) | 8.67 (4.70) | 8.37 (6.59)
  Change at Week 12 | 4.09 (5.03) | 10.21 (4.86) | 18.47 (10.06)
  Change at Week 18 | 8.14 (5.16) | 12.29 (4.93) | 11.30 (13.70)
  Change at Week 24 | 9.86 (5.42) | 9.70 (5.09) | -0.15 (13.71)
  Change at Week 30 | 9.09 (5.38) | 13.84 (5.11) | 6.88 (13.71)
  Change at Week 36 | 9.18 (5.49) | 17.49 (5.16) | -3.20 (16.31)
  Change at Week 42 | 8.15 (5.62) | 14.01 (5.26) | 29.87 (16.32)
  Change at Week 48 | 12.04 (5.63) | 16.09 (5.26) | 6.36 (16.33)

13. Secondary Outcome: Participant Pain Visual Analog Scale (VAS) at Randomization
Description: Participants indicated the amount of pain experience during the last 2-3 days by marking a vertical line on 100 mm VAS. Intensity of pain range: 0 = no pain to 100 = pain as bad as it could be.
Time Frame: Randomization (Week 0)
Population: m-ITT analysis set.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
mm | 15.59 (18.16) | 12.96 (10.92) | 13.37 (10.05)

14. Secondary Outcome: Change From Randomization in Participant Pain Visual Analog Scale (VAS) at Week 6, 12, 18, 24, 30, 36, 42, and 48
Description: as for outcome 13
Time Frame: Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: m-ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
mm
  Change at Week 6 | 1.90 (3.32) | 5.67 (3.69) | 22.70 (6.39)
  Change at Week 12 | -3.05 (3.56) | 8.05 (3.84) | 34.27 (9.43)
  Change at Week 18 | 2.21 (3.61) | 12.21 (3.90) | 12.91 (12.40)
  Change at Week 24 | -1.18 (3.88) | 7.46 (4.06) | 11.32 (12.41)
  Change at Week 30 | 3.20 (3.81) | 7.13 (4.08) | 15.97 (12.41)
  Change at Week 36 | 2.05 (3.90) | 13.00 (4.15) | 1.46 (14.49)
  Change at Week 42 | 1.06 (4.02) | 12.84 (4.26) | 7.13 (14.49)
  Change at Week 48 | 1.32 (4.06) | 9.13 (4.28) | 6.47 (14.50)

15. Secondary Outcome: Change From Randomization in Morning Stiffness Duration at Week 6, 12, 18, 24, 30, 36, 42, and 48
Description: Duration of morning stiffness: Time elapsed when participant woke up in morning and was able to resume normal activities without stiffness in minutes. The duration of morning stiffness was determined by asking the following questions: 1) Over the last 2 days, when did you wake in the morning? 2) Over the last 2 days, when were you able to resume your normal activities without stiffness? Increase in stiffness duration from randomization represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: as for outcome 9
Measure: Median (Full Range); unit: minutes
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 26 | 23
minutes
  Randomization (n=23,26,23) | 10.0 [0 to 240] | 0.5 [0 to 240] | 5.0 [0 to 120]
  Change at Week 6 (n= 22, 25, 15) | 0.0 [-60 to 50] | 0.0 [-30 to 120] | 0.0 [-5 to 1440]
  Change at Week 12 (n= 18, 20, 5) | 0.0 [-15 to 10] | 0.0 [-30 to 1410] | 1.0 [0 to 60]
  Change at Week 18 (n= 16, 19, 3) | 0.0 [0 to 1410] | 0.0 [-30 to 1410] | 0.0 [-5 to 15]
  Change at Week 24 (n= 14, 16, 3) | 0.0 [-30 to 5] | 0.0 [-60 to 90] | 0.0 [-5 to 0]
  Change at Week 30 (n= 14, 15, 3) | 0.0 [-15 to 330] | 0.0 [-110 to 60] | -5.0 [-15 to 0]
  Change at Week 36 (n= 13, 14, 2) | 0.0 [-15 to 0] | 0.0 [-120 to 60] | -2.5 [-5 to 0]
  Change at Week 42 (n= 12, 11, 2) | 0.0 [-10 to 5] | 0.0 [-120 to 60] | -2.5 [-5 to 0]
  Change at Week 48 (n= 12, 11, 2) | 0.0 [-10 to 15] | 0.0 [-30 to 60] | -5.0 [-10 to 0]

16. Secondary Outcome: Change From Randomization in Erythrocyte Sedimentation Rate (ESR) at Week 6, 12, 18, 24, 30, 36, 42, and 48
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeter per hour (mm/hour). A higher rate is consistent with inflammation.
Time Frame: Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: as for outcome 9
Measure: Median (Full Range); unit: mm/hour
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 22 | 27 | 23
mm/hour
  Randomization (n=22,27,23) | 10.00 [2.0 to 30.0] | 8.00 [1.0 to 22.0] | 8.00 [1.0 to 20.0]
  Change at Week 6 (n= 21, 26, 15) | 0.00 [-8.0 to 10.0] | 0.00 [-14.0 to 26.0] | 2.00 [-6.0 to 26.0]
  Change at Week 12 (n= 17, 21, 6) | 0.00 [-7.0 to 15.0] | 0.00 [-8.0 to 11.0] | 0.50 [-8.0 to 7.0]
  Change at Week 18 (n= 15, 19, 3) | 1.00 [-6.0 to 25.0] | 1.00 [-7.0 to 32.0] | 2.00 [-6.0 to 10.0]
  Change at Week 24 (n= 14, 16, 3) | -1.00 [-14.0 to 10.0] | 0.00 [-5.0 to 21.0] | 1.00 [-6.0 to 4.0]
  Change at Week 30 (n= 14, 15, 3) | -1.50 [-15.0 to 23.0] | 0.00 [-4.0 to 27.0] | 1.00 [-4.0 to 5.0]
  Change at Week 36 (n= 13, 14, 2) | 0.00 [-7.0 to 4.0] | 1.50 [-5.0 to 45.0] | -2.50 [-6.0 to 1.0]
  Change at Week 42 (n= 12, 12, 2) | -1.50 [-14.0 to 1.0] | 0.00 [-7.0 to 11.0] | -0.50 [-4.0 to 3.0]
  Change at Week 48 (n= 12, 12, 2) | 2.00 [-4.0 to 36.0] | 1.00 [-3.0 to 43.0] | -2.50 [-6.0 to 1.0]

17. Secondary Outcome: Change From Randomization in C-Reactive Protein (CRP) Level at Week 6, 12, 18, 24, 30, 36, 42, and 48
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range of CRP is <10 milligram per liter (mg/L). A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Randomization (Week 0), Week 6, 12, 18, 24, 30, 36, 42, 48
Population: m-ITT analysis set. Here, 'n' signifies participants evaluable for each time point for each treatment arm, respectively.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
mg/L
  Randomization (n=23,27,23) | 2.00 [0.6 to 12.0] | 3.00 [0.2 to 66.0] | 1.60 [0.6 to 8.0]
  Change at Week 6 (n= 22, 26, 15) | 0.00 [-9.0 to 59.0] | 0.00 [-33.2 to 31.7] | 0.33 [-3.0 to 17.9]
  Change at Week 12 (n= 18, 20, 6) | 0.00 [-10.0 to 44.0] | 0.00 [-63.4 to 12.0] | 0.00 [-3.0 to 4.1]
  Change at Week 18 (n= 16, 19, 3) | 0.00 [-4.0 to 12.0] | 0.00 [-4.0 to 139.0] | 2.74 [1.0 to 26.4]
  Change at Week 24 (n= 14, 16, 3) | 0.00 [-4.0 to 1.1] | 0.00 [-3.1 to 2.5] | 1.00 [0.2 to 4.3]
  Change at Week 30 (n= 14, 15, 3) | 0.00 [-3.0 to 5.1] | 0.00 [-3.0 to 9.0] | 1.20 [1.0 to 73.6]
  Change at Week 36 (n= 13, 14, 2) | 0.00 [-2.0 to 2.9] | 0.00 [-5.0 to 29.8] | 0.94 [0.0 to 1.9]
  Change at Week 42 (n= 12, 12, 2) | 0.00 [-3.0 to 1.0] | 0.00 [-3.1 to 1.0] | 3.49 [3.0 to 4.0]
  Change at Week 48 (n= 12, 12, 2) | 0.00 [-4.0 to 45.0] | 0.00 [-5.0 to 6.0] | -1.42 [-3.8 to 1.0]

18. Secondary Outcome: Change From Randomization in Modified Total Sharp Score (mTSS) at Week 48
Description: mTSS = sum of erosion and Joint Space Narrowing (JSN) scores for 44 joints (16 per hand and 6 per foot). mTSS scores ranged from 0 (normal) to 448 (worst possible total score). Change: scores at observation minus score at randomization. An increase in mTSS from randomization represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Randomization (Week 0), Week 48
Population: as for outcome 9
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 19 | 22 | 17
units on a scale
  Randomization (n=19, 22, 17) | 19.50 [0.5 to 176.0] | 54.25 [3.5 to 219.0] | 23.00 [4.0 to 89.5]
  Change at Week 48 (n= 9, 9, 1) | 0.00 [-1.0 to 0.0] | 0.00 [-2.0 to 0.5] | -1.00 [-1.0 to -1.0]

19. Secondary Outcome: Magnetic Resonance Imaging (MRI) Findings at Randomization
Description: MRI of hand/wrist of dominant hand scored for signs of synovitis (S-score), bone edema(O-score), bone erosions (E-score) as per outcome measures in RA clinical trials (OMERACT). S-score:0(normal)-3(severe) for distal radioulnar,radiocarpal,intercarpal-carpometacarpal,second-fifth metacarpophalangeal joints, total score(TS)0-21, higher score(HS)=severe synovitis. O-score:0(no volume increment)-3(100% volume increment) in 23 hand/wrist joints, TS 0-69, HS=more edema. E-score:0(no volume occupied by erosion)-10(100% volume occupied by erosion) in 23 hand/wrist joints, TS 0-230, HS=more erosion.
Time Frame: Randomization (Week 0)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 18 | 21 | 15
units on a scale
  S-Score | 4.19 (3.13) | 4.90 (3.26) | 4.37 (4.43)
  O-Score | 1.50 (1.34) | 3.14 (3.95) | 3.63 (3.36)
  E-Score | 12.53 (18.47) | 25.10 (28.23) | 12.60 (10.80)

20. Secondary Outcome: Change From Randomization in Magnetic Resonance Imaging (MRI) Findings (S-Score) at Week 12
Description: MRI of hand/wrist of dominant hand was scored for signs of synovitis (S-score), bone edema (O-score), and bone erosions (E-score) as per OMERACT. S-score: 0 (normal) to 3 (severe) for each of distal radioulnar, radiocarpal, intercarpal-carpometacarpal, second to fifth metacarpophalangeal joints; total score 0 to 21, higher score=severe synovitis.
Time Frame: Randomization (Week 0), Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 15 | 14 | 3
units on a scale | -0.16 (0.56) | 1.36 (0.68) | -0.29 (1.15)

21. Secondary Outcome: Change From Randomization in Magnetic Resonance Imaging (MRI) Findings (O-Score, E-Score) at Week 12
Description: MRI of hand/wrist of dominant hand was scored for signs of synovitis (S-score), bone edema (O-score), and bone erosions (E-score) as per OMERACT. O-score: 0 (no volume increment) to 3 (100% volume increment) in 23 hand/wrist joints; total score 0 to 69, higher scores=more edema. E-score: 0 (no volume occupied by erosion) to 10 (100% volume occupied by erosion) in 23 hand/wrist joints; total score 0 to 230, higher scores=more erosion.
Time Frame: Randomization (Week 0), Week 12
Population: as for outcome 4
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 15 | 14 | 3
units on a scale
  Change at Week 12: O-Score | 0.00 [-2.0 to 0.0] | 0.00 [-0.5 to 2.0] | -3.00 [-4.0 to 0.5]
  Change at Week 12: E-Score | 0.00 [-1.0 to 0.5] | 0.00 [-0.5 to 4.0] | 0.00 [0.0 to 0.0]

22. Secondary Outcome: Percentage of Participants in Treatment Failure for Each Potentially Predictor Variable at Randomization
Description: Percentage of participants who were treatment failure over 48 weeks as per potentially predictor variables (at randomization) are reported: number of swollen joints/tender joints, DAS28, PGA, PtGA, participant general health VAS, participant pain VAS, clinical disease activity index (CDAI), simplified disease activity index (SDAI), ESR (mm/hour), plasma CRP (mg/L), sensitive serum CRP (mg/L), anti- cyclic citrullinated peptide (anti CCP, units/mL), cartilage oligomeric matrix protein (COMP, units/liter), S-score, O-score, E-score, Joint space narrowing score, erosion score, and mTSS.
Time Frame: Randomization (Week 0) up to Week 48
Population: m-ITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2
Number analyzed (Participants) | 23 | 27 | 23
percentage of participants
  Number of swollen joints = 0 (n= 18, 21, 19) | 44.4 | 57.1 | 84.2
  Number of swollen joints >0 (n= 5, 6, 4) | 60.0 | 50.0 | 100
  Number of tender joints = 0 (n= 20, 19, 15) | 45.0 | 47.4 | 86.7
  Number of tender joints >0 to 1 (n= 2, 4, 6) | 100 | 75.0 | 83.3
  Number of tender joints > 1 (n= 0, 4, 2) | 0.0 | 75.0 | 100
  DAS28 <=2.6 (n= 20, 21, 18) | 40.0 | 47.6 | 83.3
  DAS28 >2.6 to 3.2 (n= 2, 5, 5) | 100 | 80.0 | 100
  DAS28 >3.2 to 5.1 (n= 0, 1, 0) | 0.0 | 100 | 0.0
  PGA = 0 (n= 6, 4, 9) | 50.0 | 25.0 | 88.9
  PGA >0 to 3 (n= 5, 10, 3) | 60.0 | 60.0 | 100
  PGA >3 to 7 (n= 9, 5, 5) | 33.3 | 40.0 | 80.0
  PGA >7 (n= 3, 8, 5) | 66.7 | 75.0 | 80.0
  PtGA <= 2.5 (n= 6, 8, 5) | 66.7 | 37.5 | 100
  PtGA >2.5 to 11 (n= 7, 5, 6) | 28.6 | 60.0 | 83.3
  PtGA >11 to 21 (n= 4, 7, 7) | 50.0 | 57.1 | 85.7
  PtGA >21 (n= 6, 7, 5) | 50.0 | 71.4 | 80.0
  Participant general health VAS <=3 (n= 6, 7, 6) | 50.0 | 28.6 | 83.3
  Participant general health VAS >3 to 14 (n= 9,8,4) | 44.4 | 62.5 | 100
  Participant general health VAS>14 to 26.5(n=2,7,7) | 100 | 57.1 | 71.4
  Participant general health VAS >26.5 (n= 6, 5, 6) | 33.3 | 80.0 | 100
  Participant pain VAS <=3 (n= 7, 8, 5) | 57.1 | 37.5 | 100
  Participant pain VAS >3 to 10 (n= 6, 5, 6) | 33.3 | 20.0 | 83.3
  Participant pain VAS >10 to 22 (n=3, 7, 8) | 33.3 | 85.7 | 87.5
  Participant pain VAS >22 (n= 7, 7, 4) | 57.1 | 71.4 | 75.0
  CDAI <= 2.8 (n= 14, 13, 13) | 50.0 | 46.2 | 84.6
  CDAI >2.8 to 10 (n= 9, 14, 9) | 44.4 | 64.3 | 88.9
  SDAI<= 3.3 (n= 8, 7, 8) | 50.0 | 28.6 | 75.0
  SDAI>3.3 to 11 (n= 13, 15, 12) | 38.5 | 60.0 | 100
  SDAI>11 to 26 (n= 2, 4, 2) | 100 | 75.0 | 50.0
  SDAI>26 (n= 0, 1, 0) | 0.0 | 100 | 0.0
  ESR<= 5 (n= 6, 8, 10) | 66.7 | 12.5 | 80.0
  ESR >5 to 10 (n= 7, 9, 6) | 28.6 | 66.7 | 100
  ESR >10 to 12.5 (n= 0, 3, 2) | 0.0 | 100 | 100
  ESR >12.5 (n= 6, 7, 5) | 66.7 | 71.4 | 80.0
  Plasma CRP <= 1 (n= 8, 8, 8) | 62.5 | 37.5 | 75.0
  Plasma CRP >1 to 2 (n= 5, 2, 7) | 20.0 | 50.0 | 100
  Plasma CRP >2 to 5 (n= 6, 11, 3) | 16.7 | 54.5 | 100
  Plasma CRP >5 (n= 4, 6, 5) | 100 | 83.3 | 80.0
  Sensitive serum CRP <= 0.6 (n= 7, 5, 6) | 57.1 | 20.0 | 83.3
  Sensitive serum CRP >0.6 to 1.2 (n= 5, 5, 7) | 40.0 | 80.0 | 85.7
  Sensitive serum CRP >1.2 to 3.3 (n= 6, 7, 5) | 33.3 | 42.9 | 100
  Sensitive serum CRP >3.3 (n= 4, 8, 5) | 75.0 | 75.0 | 80.0
  Anti-CCP <= 31.7 (n= 5, 8, 5) | 40.0 | 37.5 | 100
  Anti-CCP >31.7 to 346.8 (n= 8, 3, 6) | 75.0 | 100 | 83.3
  Anti-CCP >346.8 to 710.8 (n= 5, 4, 9) | 20.0 | 50.0 | 77.8
  Anti-CCP >710.8 (n= 4, 10, 3) | 50.0 | 60.0 | 100
  COMP <= 7.6 (n= 7, 5, 6) | 28.6 | 20.0 | 66.7
  COMP >7.6 to 9.6 (n= 5, 4, 8) | 60.0 | 50.0 | 100
  COMP >9.6 to 12.3 (n= 5, 11, 2) | 80.0 | 63.6 | 100
  COMP >12.3 (n= 5, 5, 7) | 40.0 | 80.0 | 85.7
  S-score <= 1.5 (n= 5, 5, 5) | 20.0 | 40.0 | 80.0
  S-score >1.5 to 3.8 (n= 5, 2, 5) | 20.0 | 50.0 | 60.0
  S-score >3.8 to 7.5 (n= 5, 8, 1) | 80.0 | 37.5 | 100
  S-score >7.5 (n= 3, 6, 4) | 66.7 | 50.0 | 100
  O-score <= 0.5 (n= 6, 7, 4) | 16.7 | 42.9 | 50.0
  O-score >0.5 to 1.5 (n= 4, 6, 2) | 25.0 | 50.0 | 100
  O-score >1.5 to 3.5 (n= 7, 0, 3) | 71.4 | 0.0 | 100
  O-score >3.5 (n= 1, 6, 6) | 100 | 50.0 | 83.3
  E-score <= 3.0 (n= 7, 5, 5) | 14.3 | 20.0 | 60.0
  E-score >3.0 to 9.8 (n= 4, 4, 2) | 75.0 | 25.0 | 100
  E-score >9.8 to 23.0 (n= 5, 4, 5) | 60.0 | 50.0 | 80.0
  E-score >23.0 (n= 2, 8, 3) | 50.0 | 62.5 | 100
  Joint space narrowing score <= 0.5 (n= 5, 7, 5) | 20.0 | 28.6 | 60.0
  Joint space narrowing score >0.5 to 9.0 (n=5,0,6) | 60.0 | 0.0 | 100
  Joint space narrowing score >9.0 to 23.5 (n=7,4,3) | 57.1 | 75.0 | 66.7
  Joint space narrowing score >23.5 (n= 2, 9, 3) | 50.0 | 66.7 | 100
  Erosion score <= 9.0 (n= 7, 0, 3) | 42.9 | 0.0 | 66.7
  Erosion score >9.0 to 21.3 (n= 4, 3, 7) | 25.0 | 66.7 | 85.7
  Erosion score >21.3 to 47.5 (n= 5, 6, 4) | 40.0 | 50.0 | 75.0
  Erosion score >47.5 (n= 3, 8, 3) | 100 | 75.0 | 100
  mTSS <= 10.0 (n= 5, 6, 4) | 20.0 | 16.7 | 50.0
  mTSS >10.0 to 31.5 (n= 5, 3, 6) | 60.0 | 33.3 | 100
  mTSS >31.5 to 70.0 (n= 7, 4, 4) | 42.9 | 75.0 | 75.0
  mTSS >70.0 (n= 2, 9, 3) | 100 | 66.7 | 100

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept 50 mg - Period 1 | Etanercept 50 mg - Period 2 | Etanercept 25 mg - Period 2 | Placebo - Period 2 | Etanercept 50 mg - Period 3
Serious Adverse Events (participants affected / at risk) | 0/91 | 1/23 | 1/27 | 0/23 | 1/43
Other Adverse Events (participants affected / at risk) | 27/91 | 16/23 | 20/27 | 7/23 | 31/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept 50 mg - Period 1 (N=91) | Etanercept 50 mg - Period 2 (N=23) | Etanercept 25 mg - Period 2 (N=27) | Placebo - Period 2 (N=23) | Etanercept 50 mg - Period 3 (N=43)
Endometritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept 50 mg - Period 1 (N=91) | Etanercept 50 mg - Period 2 (N=23) | Etanercept 25 mg - Period 2 (N=27) | Placebo - Period 2 (N=23) | Etanercept 50 mg - Period 3 (N=43)
Nasopharyngitis (Infections and infestations) | 7 | 6 | 8 | 2 | 8
Upper respiratory tract infection (Infections and infestations) | 2 | 6 | 3 | 2 | 9
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 0 | 3
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Erythema migrans (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Borrelia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Enterobiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 3 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 3 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1
Dental operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Toe operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Photokeratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Benign neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.